CLINICAL TRIAL: NCT06772142
Title: Early Feasibility of the Nervonik Peripheral Nerve Stimulation Device
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Nervonik (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CIP 001
Record Dates: First submitted 2024-12-27; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Peripheral Nerve Disorder
Keywords: peripheral; nerve; stimulation
MeSH Terms: conditions — Neuritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (2):
- COHORT 1, Acute (Other): The initial cohort of patients will receive the Nervonik neurostimulator for up to 8 hours. The patient will remain local to the care facility for implant stimulator program changes until the patient is satisfied with the degree of pain relief. The implant will be removed from the patient at the end of the evaluation.
  Interventions: Device: Peripheral Nerve Stimulation
- COHORT 2, Chronic (Other): The second cohort of patients will include those patients from cohort 1 who have determined the Nervonik implant provides suitable pain relief and agree to have a permanent implant placed. In addition, the second cohort includes non-cohort one patients meeting the trial requirements and agreeing to participate in the trial.
  Interventions: Device: Peripheral Nerve Stimulation

INTERVENTIONS:
Device: Peripheral Nerve Stimulation — Peripheral Nerve Stimulation

SUMMARY:
A multicenter, 30 patient prospective single arm evaluation of the Nervonik system in symptomatic patients with chronic severe knee, elbow or shoulder pain.

COHORT 1: The initial cohort of patients will receive the Nervonik neurostimulator for up to 8 hours. The patient will remain local to the care facility for implant stimulator program changes until the patient is satisfied with the degree of pain relief. The implant will be removed from the patient at the end of the evaluation.

COHORT 2: The second cohort of patients will include those patients from cohort 1 who have determined the Nervonik implant provides suitable pain relief and agree to have a permanent implant placed. In addition, the second cohort includes non-cohort one patients meeting the trial requirements and agreeing to participate in the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is between 18 to 80 years of age at the time of enrollment.
2. Subject has been diagnosed with knee, arm, or shoulder chronic pain (NRS of at least 5 out of 10).
3. Post-surgical/post-traumatic peripheral neuralgia including but not limited to pain due to peripheral nerve injury, post-surgical scar formation, nerve entrapment; Mononeuropathy, specified or unspecified or in diseases classified elsewhere; Other neuralgia or neuropathic pain
4. Subject is willing to cooperate with the study requirements including, compliance with the study procedures and completion of all study visits.
5. Subject reported stable pain (non-escalating) for 60 days prior to signing informed consent.
6. Subject is currently receiving CMM and has had stable pain medication use and dosage for 30 days prior to signing informed consent.
7. Subject is psychologically qualified to receive a peripheral nerve stimulator as per the clinician's standard clinical practice and judgment and does not have clinically relevant psychological condition(s) that would interfere with their ability to accurately report outcomes or complete study procedures.
8. Subject has demonstrated the ability to appropriately place the wearable in the location where the IPG is most likely to be implanted. Alternatively, subject is able to appropriately use the relief belt and/or limb cuff to keep the wearable in place.

Exclusion Criteria:

1. Subject currently has an active implantable medical device such as a drug pump, spinal cord stimulator, peripheral nerve stimulator, sacral nerve stimulator, deep brain stimulator, and/or cardiac pacemaker.
2. Subject has previously failed PNS or Spinal Cord Stimulation (SCS) or Dorsal Root Ganglion (DRG) therapy (trial or permanent implant). See note below.
3. Pain is completely absent at rest.
4. Patient has clinical evidence of complex regional pain syndrome (CRPS), peripheral neuralgia of metabolic origin, post-herpetic neuralgia, biochemical evidence of a metabolic or genetic neuropathy (e.g., Charcot'- Marie- Tooth Disease) or mixed motor/sensory polyneuropathy.
5. Subject has a medical condition that would prevent them from participating in the current study per investigator's or medical monitor's judgment.
6. Subject has had a successful (≥ 50% pain relief) interventional procedure within the past 3 months to treat the same pain condition(s) being examined in this study including, nerve blocks.
7. Uncontrolled depression or uncontrolled psychiatric disorders
8. Subject is currently participating in another clinical investigation with an active treatment arm.
9. Subject is allergic or sensitive to materials used in the device components including, skin adhesives or does not tolerate the wearable aspect of the device.
10. Subject has pending or ongoing legal issues (including unresolved worker's compensation claims or equivalent) or other conflicting secondary gain issues related to their chronic pain condition.
11. Subject has a current diagnosis of a coagulation disorder, bleeding diathesis, or progressive peripheral vascular disease that has not been medically corrected.
12. Subject has an active systemic infection.
13. Subject is unable to read and/or write in Spanish or give informed consent.
14. Subject has a life expectancy of less than 1 year
15. Subject has an active malignant neoplasm (metastatic or local) or evidence of paraneoplastic syndrome.
16. Subject with uncontrolled diabetes mellitus, showing signs of diabetic neuropathy, as evidenced by a neurological exam and a HbA1c test.
17. Subject has evidence of an alcohol or drug dependency within the last 6 months prior to enrollment.
18. Subject is pregnant (if female and sexually active, subject must be using a reliable form of birth control, be surgically sterile or be at least 1 year post-menopausal).
19. Subject is nursing/breastfeeding.
20. Subject is on ≥90 mg-morphine equivalents per 24 hours. Recommend 60.
21. Subject has undergone an ablative treatment of the target peripheral nerve, or proximal nerve trunk giving rise to the target nerve, or dorsal roots (and DRGs) that ultimately make up the target nerve. No ablative procedures directed at the spinal cord, dorsal roots, or peripheral nerve(s) being treated in the study. To note, subjects who have undergone RF ablation of the dorsal rami, cool pulsed RF of the facet innervation may be considered for enrollment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint 1 | Through study completion, average of 1 day [Cohort 1] and average of 1 year [Cohort 2]
  Safety - reporting of adverse events
Primary Endpoint 2 | Through study completion, average of 1 day [Cohort 1] and average of 1 year [Cohort 2]
  Device performance - successfully delivering current to the nerve

SECONDARY OUTCOMES:
Secondary Outcome 1 | Through study completion, average of 1 day [Cohort 1] and average of 1 year [Cohort 2]
  Average pain intensity, Long Term durability of Average Pain Intensity (Numeric Rating Scale (NRS)
Secondary Outcome 2 | Through study completion, average of 1 day [Cohort 1] and average of 1 year [Cohort 2]
  Patient Global Impression of Change (PGIC) - PGIC assesses the patient's impression of change in quality of life.
Secondary Outcome 3 | Through study completion, average of 1 day [Cohort 1] and average of 1 year [Cohort 2]
  Patient Interview

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Punta Pacifica, Panama City, Provincia de Panamá, Panama